CLINICAL TRIAL: NCT01348763
Title: A Phase 1 Pharmacokinetic Study to Assess the Steady State Pharmacokinetic Profile and Short Term Safety of Maraviroc Dosed With Darunavir/Ritonavir All Once Daily, With and Without Nucleoside Analogues, in HIV-1 Infected Subjects
Brief Title: The Maraviroc Darunavir/Ritonavir Once Daily Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MRV_DRV_PK; 2009-014924-42 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-05-05 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: HIV
MeSH Terms: interventions — Maraviroc; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Truvada, Darunavir/r and Maraviroc (Experimental): Participants will be taking Truvada, Darunavir/r before entering the study. On day 1 they will add maraviroc then on day 11 they will stop the Truvada
  Interventions: Drug: Maraviroc; Drug: Truvada; Drug: Darunavir

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 150 mg daily
Drug: Truvada — daily until 10. day then stop
Drug: Darunavir — daily until 10. day then stop

SUMMARY:
This is a phase I, open label, prospective, two phase pharmacokinetic study. Subjects currently attending for HIV care at St. Mary's Hospital, London will be eligible.

DETAILED DESCRIPTION:
The study will describe the steady state pharmacokinetic parameters and short term safety of maraviroc/darunavir/ritonavir dosed at 150/800/100 mg once daily with and without tenofovir/emtricitabine 245/200 mg once daily in HIV-1 infected subjects.

Fifteen HIV-1 infected subjects will be recruited. Eligible subjects will currently be receiving antiretroviral therapy comprising:

* tenofovir/emtricitabine 245/200 mg daily plus
* darunavir/ritonavir 800/100 mg daily

On day 1, subjects will modify their current antiretroviral therapy to the following:

* tenofovir/emtricitabine 245/200 mg daily plus
* darunavir/ritonavir 800/100 mg daily plus
* maraviroc 150 mg daily On day 10 subjects will undergo an intensive pharmacokinetic visit.

On day 11, subjects will modify their current antiretroviral therapy to the following:

* darunavir/ritonavir 800/100 mg daily plus
* maraviroc 150 mg daily (i.e. tenofovir/emtricitabine will be discontinued) On day 20 subjects will undergo an intensive pharmacokinetic visit. Following completion of this study phase, subjects will recommence their usual antiretroviral treatment regimen and attend for a study follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* signed informed consent
* plasma HIV RNA < 50 copies/mL at screening and on at least one other occasion over the last 3 months
* currently receiving an antiretroviral regimen comprising of: tenofovir 245 mg daily,emtricitabine 200 mg daily, darunavir 800 mg daily and ritonavir 100 mg daily
* no previous protease inhibitor resistance documented on HIV-1 genotypic resistance testing if an HIV resistance test available
* Between 18 to 65 years of age, inclusive
* subjects in good health upon medical history, physical exam, and laboratory testing
* BMI above or equal to 18 and below 32
* Female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must practice contraception as follows from screening until 8 weeks after completion of the study:
* barrier contraceptives (condom OR diaphragm PLUS spermicide) or oral, implant or injectable hormonal contraceptive PLUS a barrier contraceptive or
* IUD /IUS PLUS a barrier contraceptive
* Female subjects of childbearing potential must have a negative urine pregnancy test.
* Male subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom with spermicide) during heterosexual intercourse, from screening through completion of the study.
* Have no serologic evidence of active HBV infection evidenced by negative hepatitis B surface antigen and no serologic evidence of hepatitis C virus infection evidenced by a negative HCV antibody at screening.
* Have screening laboratory results (haematology and chemistry that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance
* CCR5 tropic HIV virus based on a genotypic tropism assay from either a stored plasma sample where available or fresh plasma

Exclusion Criteria:

* current alcohol abuse or drug dependence
* positive urine drug of abuse screening
* pregnancy
* active opportunistic infection or significant co-morbidities
* current disallowed concomitant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male only
Enrollment: 13 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MB BH, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mora-Peris B, Croucher A, Else LJ, Vera JH, Khoo S, Scullard G, Back D, Winston A. Pharmacokinetic profile and safety of 150 mg of maraviroc dosed with 800/100 mg of darunavir/ritonavir all once daily, with and without nucleoside analogues, in HIV-infected subjects. J Antimicrob Chemother. 2013 Jun;68(6):1348-53. doi: 10.1093/jac/dkt006. Epub 2013 Jan 30. PMID 23364475

RESULTS

PARTICIPANT FLOW:
Period: With Tenofovir/Emtricitabine (10 Days)
Arm/Group | Truvada, Darunavir/r and Maraviroc
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: Without Tenofovir/Emtricitabine (11 Day)
Arm/Group | Truvada, Darunavir/r and Maraviroc
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Truvada, Darunavir/r and Maraviroc
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: The Ratio of the Maximum Plasma Concentration of Maraviroc Between 20 and 10 Day
Description: On day 10 of the study the maximum concentractions of maraviroc will be measured . On day 20 of the study the maximum plasma concentractions maraviroc will be measured .
Time Frame: 10 day, 20 days
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Truvada, Darunavir/r and Maraviroc
Number analyzed (Participants) | 11
ratio | 0.99 [0.79 to 1.25]

2. Secondary Outcome: Number of Participants With Changes in Haematology and Biochemistry Laboratory Tests
Description: Haematology and biochemistry laboratory tests such as full blood count, elelectrolytes and lipids will be measured to assess for changes.
Time Frame: 35 days
Population: No data reported
Measure: Count of Participants; unit: Participants
Arm/Group | Truvada, Darunavir/r and Maraviroc
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Truvada, Darunavir/r and Maraviroc
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes